CLINICAL TRIAL: NCT05362435
Title: Expansion and Spread of Makoyoh'Sokoi, the Wolf Trail, a Community Led, Culturally Relevant, Physical Activity-based, Holistic Wellness Program for Indigenous Women; a Self-control, Non- Randomized, Intervention Trial in Seven Communities (10 Sites) in Alberta and Saskatchewan
Brief Title: Makoyoh'Sokoi - The Wolf Trail Program Expansion Project - Supporting Indigenous Women to Celebrate Good Health
Acronym: MKS+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-1305
Record Dates: First submitted 2022-02-22; First posted 2022-05-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This will be a self-control, non-randomised intervention. Participant data collection will occur at the following times:
  Cohort A & B T1 = 3 months pre-program T2 = Week 1 = immediately pre-program T3 = Week 12 = post live program (12 weeks) T4 = Week 24 = post full program T5 = 1 year after T4
  Cohort C, D, E 3-month control removed after consultation. T1 = Week 1 = immediately pre-program T2 = Week 12 = post live program (12 weeks) T3 = Week 18 or 24 = post full program T4 = 1 year after T4
  Data input will occur in March and July annually, there will be 5 cohorts over the three years (Jan 2022 [COHORT A], Sept 2022 [COHORT B], Jan 2023 [COHORT C], Sept 2023 [COHORT D], Jan 2024 [COHORT E]). Cohorts A, B, C will have all data points collected, cohorts D and E will not have data collected 1-year post completion (unless the researchers are able to extend funding to include the one-year follow-up for these cohorts). Each cohort will be exposed to the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participation in Makoyoh'sokoi (the Wolf Trail Program) (Experimental): This is a self-control, non-randomised intervention study. 7 locations will run a total of 10 programs (4 urban, off-reserve; 6 rural, on reserve).
  Makoyoh'sokoi (The Wolf Trail Program) is a holistic health and wellness program that consists of a 12-week live phase where participants engage weekly in approximately 45 minutes of physical activity, 20 minutes of a health education module, and 20 minutes of a sharing circle. The live phase is followed by a 12-week follow-up phase where participants meet bi-weekly for approximately 30 minutes of a health education module and 30 minutes of a sharing circle.
  Interventions: Behavioral: Physical activity-based wellness programs

INTERVENTIONS:
Behavioral: Physical activity-based wellness programs — Each MKS+ program has 20-25 participants and consists of the following: 12 Week INTENSE PHASE: 1) pre-program information and orientation session, and data collection/testing; 2) core weekly programming with the following three components: a) 45-60 minute exercise class, b) 15-20 minute nutrition and wellness education, and c) 15-30 minute sharing circle; 3) end of program celebration; 4) urban poling sessions; 5) introduction to local healthcare providers as identified as relevant for the group; 6) ongoing online support via private Facebook group; 7) daily pedometer tracking to provide immediate motivational feedback to participants. 6-12 Week FOLLOW-UP PHASE: 1) Program Facilitator contacts participants weekly to encourage healthy activities, address concerns as needed, and record weekly step counts; 2) encourages continued engagement in private Facebook group; 3) 15-30 minute nutrition and wellness education, and c) 15-45 minute sharing circle.

SUMMARY:
During the MKS+ program participants complete health education modules that expose them to health information, a substantial portion of which relate to healthy nutrition and prevention, and on occasion to local healthcare providers. The goal is to increase activation and the ability to manage one's own health. In each community, the Community Organisational Leads will support the Facilitators to establish a comprehensive resource list of healthcare professionals. Additionally, through exposure to local Indigenous Knowledge Keepers and Elders, along with cultural and spiritual elements, the participants will know how to access activities that may further support their wellness. The MKS+ program shows promise as a community-based model for supporting Indigenous women to improve their health. It is grounded in community; increases self-efficacy through the opportunity to learn, practice, and share in manageable increments; and increases health literacy through program contents and coordinating healthcare knowledge exchange with other healthcare providers from the community. By connecting to aspects of Indigenous culture, participants can be affirmed in their identities and learn more about how connecting to culture may be protective of their health through a restored sense of self-worth, sharing, and community support.

At the individual participant level the investigators anticipate the participants will a) improve their fitness, body composition and cardiometabolic health, b) improve their quality of life and mental health, c) develop strong support networks, d) be exposed to cultural elements in their community that the participants were not previously aware of that may lead to engagement, better understanding and easier access to their community resources, e) learn about healthy diet composition - shopping, cooking, and meal planning which will lead to improved nutrition, and f) understand the importance of health screening and smoking cessation. The investigators' earlier pilot work established these outcomes and the investigators are hopeful because this project will support an extended program that will include an additional 12 weeks of less intense, follow-up programming, that the investigators will also find that these elements are sustained at one-year post-programming. In previous grants, the investigators have never had the opportunity to extend the program in this way.

DETAILED DESCRIPTION:
The Makoyoh'sokoi (Wolf Trail) Program is a holistic wellness program that is highly integrated both in its capacity as a program and in its mission to support its participants. In doing so the program has multiple areas of evaluation. The focus of the program evaluation is on making the evaluative measurements meaningful to either the participants or the community. The evaluative elements will be woven into the education components of the program so that each element/result is presented to a participant in such a way that it is meaningful to them and will assist them in their health journey. All elements not directly meaningful to either participants or the community have been reviewed, justified and agreed upon by community leads.

Participants will be women of all ages, 18 and older. The benefit of being inclusive of all ages is that there is intergenerational knowledge sharing and support, and role modelling can occur. In previous programs having a wide range of ages was always seen as a benefit for this reason and not as a deficit, despite the varied abilities to perform the physical exercise. To deal with the latter, the fitness instructors are well versed on adapting the exercises to the participants based on ability. An evaluation of the role of past participants from Lloydminster revealed that, on average, the program participants were responsible for food, clothing and care of 7-8 individuals each (research by Megan Sampson, Master's student), many caring for multiple generations and multiple families. The age of participants in all previous programming varied, the means ranged from 37-39 years old.

As this is a self-control, non-randomised study, with an evaluative component, no pre-set power calculations were made. Sample size is based largely on the size of the room available to host the classes along with the budget and available in-kind resources with a target of 25 participants initially enrolled and 20 completing each program. 25 participants will be recruited for each program, if individuals do not complete all the T1 measures then new individuals will be taken from the waiting list. If individuals drop out within the first 3 weeks, then new individuals will be taken from the waiting list. The goal will be to have 20 women complete each program. The investigators will need to define completion. The program is 24 weeks long with a total of 18 sessions.

All of the quantitative data will show descriptive statistics including mean, standard deviation (SD), or median with inter-quantile range (IQR) for continuous data and counts with percentages for categorical data. Statistical testing and modeling methods including t-test (continuous data) and chi-square test (for categorical data) will be applied to evaluate changes in key measures pre- and post programming. Nonparametric methods for example Mann-Whitney test, Kruskal-Wallis test and Mood's median test will be applied where the continuous data show significant skewness or pattern far from normal distribution. Repeated measurements ANOVA and other longitudinal models including linear mixed model or generalized linear mixed model or quantile regression (depending on outcomes' distributions) will be used to identify factors that drive the changes of key outcomes collected at T1 - T4. In addition, machine learning methods, for example, k-means clustering, regression tree or random forest, will be employed to identify subgroups with different patterns of changes in multiple outcomes through the programming. The investigators are especially interested to investigate which group(s) of patients have significant improvement in physical activities and health outcomes, and which group(s) don't have changes in outcomes. If presence of missing values and drop-outs, some inverse probability weighted likelihood methods may be used to consider the informative messiness.

All data will be collected on-site or through Qualtrics (online) for this study. The post-program data will be collected on-site also. If participants are unable to attend the class during which measurements will be completed, then the participants will be called and arrangements will be made for them to meet with the facilitator within two weeks of that date.

ELIGIBILITY:
Inclusion Criteria:

* Indigenous women from the following participating communities in rural and urban Alberta and Saskatchewan: Calgary (3 communities), Edmonton, Onion Lake Cree Nation, Waterhen Lake First Nation, Flying Dust First Nation, Ministikwan Lake Cree Nation, and Piikani Nation.
* Indigenous women may identify as Métis, First Nations or Inuit, living both on- and off-reserve
* Women, defined as gender female, and may include cis-female, binary, trans- females, queer and two-spirited individuals.
* 18 years old and older.

Exclusion Criteria:

* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women, defined as gender female, and may include cis-female, binary, trans- females, queer and two-spirited individuals.
Enrollment: 1250 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Activation | PAM scores will be collected immediately pre-program (Week 1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Participants' engagement in their own healthcare as measured by the Patient Activation Measure (PAM™). Patient activation implies a "willingness and ability to take independent actions to manage their health and care". The PAM™ score has been used to assess effectiveness of diabetes prevention programming in Indigenous populations. It is a well-validated tool to assess effectiveness of interventions for many chronic diseases and small increases in PAM score have been shown to correlate to reduced healthcare costs and improved health status. PAM™ levels are defined as follows: Level 1 <47, Level 2 47.1 - 55.1, Level 3 55.2 - 67.0, Level 4 >67.1. To assess changes in PAM™ scores over time the analysis will focus on score changes within each level. Previous studies show that most change occurs within the lowest levels of activation (Levels 1 and 2), and patients with lower activation also tend to have higher utilization and costs. So, both the PAM™ score and PAM™.
Physical Activity - Change in Step Counts | Change in step-counts will be studies between the start of the program (Week 1; Time 1), the end of the live program (Week 12; Time 2), the end of the follow-up period (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  The investigators use pedometers to track weekly step counts. Pedometers were chosen to assess physical activity because they were successfully used in the previous MKS programs, provide immediate motivational feedback to participants, and are cost effective and validated. Pedometer use will be evaluated the following ways: 1) # who are compliant with bringing their pedometers weekly and # who have kept track of their total steps, 2) average % change in weekly step count between Time 2, Time 3 and Time 4 (or last class attended) (presented as mean +/- SD, median and range). 3) % reporting continued use of their pedometer at Time 5. 4)
Physical Activity - Change in International Physical Activity Questionnaire Results | The N-IPAQ will be completed immediately pre-program (Week1; Time 1), after the live program (12 weeks; Time 2), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  The Neighbourhood - International Physical Activity Questionnaire (N-IPAQ) will be completed. The N-IPAQ is a reliable, validated, and easy to administer questionnaire that measures neighbourhood-based physical activity There are two forms of output from scoring the N-IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity. For continuous variable such as weekly step counts, MET minutes, the mean (SD) will be shown and statistical methods including paired t-test and repeated measurement ANOVA, linear (mixed effect) regression methods will be used to discover whether the program participants will have more step counts over time. For categorical data such as the level of physical activity on the N- IPAQ, the frequency distribution will be presented and Chi-square test and generalized
Participant quality of life, sense of belonging and mental health - Main | Responses will be collected immediately pre-program (Week1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Change in Mental Health Continuum-Short Form (MHC-SF) category uses three categories (languishing, moderate, flourishing) coded as 0, 1, and 2. % of participants in each category at T1, T4 and T5 will be reported along with change in category over time. Statistical method for example, two proportion test, and Chi-square tests will be used to identify whether the programming will improve the participants' well-being in three components: emotional, social, and psychological. In addition, the correlation analysis between this MHC-SF measures with other outcomes will help to reveal whether this outcome is correlated to variables such as the 12-item Short Form Survey (SF-12), Canadian Health Measures Survey GEN_18, Patient Activation Measure (PAM) and BMI (kg/m2) etc. Generalized linear mixed model will also be used for the repeated measurements collected pre and post program considering other potential factors or outcomes as adjusting covariates in the model.
Change in participant quality of life, sense of belonging and mental health - Main | Qualitative research will happen after the full program (Week 18 or 24; Time 3) and one year after the full program (Week 70 or 76; Time 4) to determine change in quality of life.
  The Medicine Wheel is a visual tool to reflect the holistic view of balance in one's life. The four quadrants are comprised of Physical, Emotional, Mental, and Spiritual. Qualitative methods will be used to explore how the program has impacted where participants are with respect to the Medicine Wheel at the end of the program, using a Medicine Wheel Likert Scale.
  A peer-researcher will be identified during the second month of each program. The peer-researcher will be trained in the photo/video-voice method. Peer-researchers will meet with participants and educate the participant on how to create a photovoice/video to answer the question. The Medicine Wheel Likert Scale is incorporated into this reflective process. The peer-researcher will support them with editing and compile the exercises.

SECONDARY OUTCOMES:
Participant cardiometabolic health - Metabolic Syndrome | Presence of metabolic syndrome will be assessed immediately pre-program (Week1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Blood pressure, waist circumference, biochemistries, and demographic data will be collected to determine prevalence of Metabolic Syndrome (MetS) and whether this changes throughout the program.
  The revised National Cholesterol Education Program Adult Treatment Panel III criteria, state that metabolic syndrome is present if three or more of the following criteria are met: abdominal obesity (waist circumference > 102 cm for men and > 88 cm for women)- numbers vary based on ethnicity; elevated plasma triglyceride level (≥ 1.7 mmol/L); decreased high-density lipoprotein (HDL) cholesterol level (< 1.03 mmol/L for men and < 1.30 mmol/L for women); elevated blood pressure (≥ 130/85 mm Hg); or elevated fasting glucose level (≥ 6.1 mmol/L).
  Report % with Met Syndrome initially for whom health improved such that they did not meet criteria at Time 4 (immediately post-program) and Time 5 (52 weeks post the end of the program).
Participant cardiometabolic health - medication usage | Medication use will be evaluated immediately pre-program (Week1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  As part of the investigators' understanding of participant cardiometabolic health, we will collect information on participant medication usage; decreasing or initiating medications for diabetes or cardiovascular risk reduction
  The descriptive statistics will be presented with mean (SD) and frequency for categorical data. The changes in those measures be analyzed by using a variety of methods such as t-test, repeated ANOVA and mixed effect model for continuous data and generalized linear mixed effect model regression for any categorized variables.
Participant cardiometabolic health - resting heart rate | Resting heart rate will be evaluated immediately pre-program (Week1; Time 1), after the live program (12 weeks; Time 2), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Resting heart rate will be evaluated as an indicator of cardiometabolic health. A lower resting heart rate at subsequent measures will be considered a sign of improved fitness. Resting heart rate is also required as part of the calculation for the 1-mile walk test.
  The descriptive statistics will be presented with mean (SD) and frequency for categorical data. The changes in those measures be analyzed by using a variety of methods such as t-test, repeated ANOVA and mixed effect model for continuous data and generalized linear mixed effect model regression for any categorized variables.
Participant cardiometabolic health - smoking status | Information on smoking status will be collected immediately pre-program (Week1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Information on smoking status, and changes to smoking status throughout the program, will be collected through a questionnaire. Reduced smoking frequency and smoking cessation will be viewed as a positive health change.
  The descriptive statistics will be presented with mean (SD) and frequency for categorical data. The changes in those measures be analyzed by using a variety of methods such as t-test, repeated ANOVA and mixed effect model for continuous data and generalized linear mixed effect model regression for any categorized variables.
Participant cardiometabolic health - CANRISK | CANRISK scores will be calculated immediately pre-program (Week1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Canadian Diabetes Risk Questionnaire (CANRISK) score
  Composed of 12 questions, CANRISK collects information on the following risk factors: age group, sex, ethnicity, education, BMI (kg/m2), waist circumference, daily physical activity, daily fruit and vegetable consumption, history of high blood pressure, blood sugar, family history of diabetes, smoking status and macrosomia.
  The CANRISK Survey evaluates diabetes risk as "low risk" (a score lower than 21), "moderate risk" (a score of 21-32), and "high risk" (a score of 33 and over).
  Report % of participants who did not have known Type-2 Diabetes Mellitus, who increased, decreased or experienced no change in CANRISK score.
Participant anthropometrics | Anthropometric measures will be completed immediately pre-program (Week1; Time 1), after the live program (12 weeks; Time 2), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Body-composition measures such as weight, height, and waist circumference will be collected, and then the investigators will calculate BMI (kg/m2), body adiposity index (BAI), and body fat percentage by using: body fat percentage= (1.20 X BMI) + 0.23 X age -5.4 (females with age >15). The data will be summarized with mean (SD) and median (IQR) for each time point at Time 1 (3 months pre-program) to Time 5 (1 year after the end of the program). The changes over time will also be evaluated by using longitudinal modeling methods (such as mixed effect model) as well as repeated measure ANOVA. The weight scale used uses impedance methods to calculate a % body fat but is limited at higher percentages. The investigators will compare percent body fat using both methods. Categorized BMI or body fat percentage based on WHO's method will be also presented with frequency and generalized linear mixed effect model will be applied to evaluate the changes over time from Time 1 to Time 5.
Fitness - Grip Strength | Grip strength will be completed immediately pre-program (Week1; Time 1), after the live program (12 weeks; Time 2), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Grip strength is found to correlate to longevity and fitness, and as participants are exposed to strength-based trainings, the investigators will use handgrip dynamometer to track the changes in strength of participants. This data will be presented with mean (SD) in different age groups and the % change from the previous time points. Linear regression will be used to evaluate whether significant changes in grip strength are observed among participants throughout and after the program the program.
Fitness - 1-mile walk test | The 1-mile walk test will be completed immediately pre-program (Week1; Time 1), after the live program (12 weeks; Time 2), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  For 1-Mile Walk Test, the data of total minutes and VO2_MAX will be calculated and presented with mean -/+ SD and the categorized data based on VO2_max are also be presented with their frequency distribution in different age groups. The changes in the measures will be evaluated based on repeated ANOVA methods and linear regression by adjusting for potential factors such as age, smoking status, BMI and so on. To perform the 1-mile walking test: 1) Warm up for 5-10 minutes. 2) Start your stopwatch and start walking as fast as you can. 3) At the end of 1 mile, record your time in decimals. 4) Take your heart rate immediately. 5) Calculate VO2_max with provided formula (VO2 max = 132.853 - (0.0769 x your weight in pounds) - (0.3877 x your age) + (6.315 if you are male or 0 if you are female) - (3.2649 x your walking time) - (0.1565 x your heart rate at the end of the test)) 6) Determine the different levels based on the provided table.
Participant quality of life, sense of belonging and mental health | EQ-5D-5L scores will be evaluated immediately pre-program (Week1; Time 1), after the live program (12 weeks; Time 2), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Improvements in quality of life will be assessed using the EQ-5D- 5L™. The investigators are going to collect three measure from EQ-5D-5L: EQ5D profile, EQ5D Vas, EQ5D measures. In addition to presenting descriptive statistics including mean (SD) and frequencies in each level for all those measures at each time points and use t-test to evaluate the changes, longitudinal analysis will be conducted to check the changes of health state before and after the intervention. Paretian Classification of Health Change (PCHC) and Health Profile Grid (HPG) will be used to summarize the change of the profile data. Linear regression models with mixed effect for both VAS and EQ5D dimension can be used to evaluate the effect of potential determinants and the effect of the programming.
Community walkability as perceived by participants | PANES scores will be will be collected immediately pre-program (Week1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  The Physical Activity Neighborhood Environment Survey (PANES) provides estimates of self- reported neighbourhood, built environment supportiveness for physical activity with some degree of test-retest reliability and construct validity. The overall PANES score should have a range of 0 to 6, with higher values indicating greater environmental support for physical activity. For each item the investigators also have a dichotomized outcome to indicate whether strongly or somewhat agree with the statement. The mean and standard deviation will be presented for the overall PANES score and percentage of participants with strongly or somewhat agree with the statement in each item. Correlations of walkability index to physical activity and fitness (and changes within these categories) will be made. Indices will be compared between sites.
Participant quality of life, sense of belonging and mental health - Secondary | Responses will be will be collected immediately pre-program (Week1; Time 1), after the live program (12 weeks; Time 2), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Social well-being will be evaluated using Canadian Health Measures Survey (CHMS) sense of belonging question: GEN_Q18: How would you describe your sense of belonging to your local community? Would you say it is?
  1. Very strong
  2. Somewhat strong
  3. Somewhat weak
  4. Very weak
  Percentage of participants in each category pre and post program will be compared and correlated with other outcome measures such as attendance, BMI, percent body fat, etc. Chi-square tests will be used to identify whether the programming will significantly change the participants' sense of belonging to their local community. Generalized linear mixed model will also be used for the repeated measurements collected pre and post program considering other potential factors such as age, income, medical history, location, education level and so on.
Participant Nutrition - Healthy Eating Index | HEI scores will be will be evaluated immediately pre-program (Week1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  The Healthy Eating Index (HEI) uses a scoring system to evaluate a set of foods. The score ranges from 0 to 100 points. The total HEI score is an indication of overall diet quality and changes in the HEI score will be used to determine whether dietary practices have improved throughout the intervention.
  Component scores when examined together show a pattern of diet quality. The summary statistics including the mean and standard deviation for the overall HEI and each component, will be included and the index value will be used as covariates when evaluating the changes in outcomes such as weight, BMI (kg/m2), PAM. Etc.
Participant Nutrition - Traditional Foods | A summary of traditional food consumption immediately pre-program (Week 1; Time 1) and after the full program (Week 18 or 24; Time 3) will be completed.
  Individual questions adapted to address Indigenous population consumption of traditional foods and changes within this category.
Participant Nutrition - Health Education | Changes in nutrition knowledge will be summarized and evaluated after the full program (Week 18 or 24; Time 3) and 52 weeks after the full program (Week 70 or 76; Time 4).
  Nutrition knowledge: Questions developed based on the Health Education Modules with a focus on nutrition elements. Questions: Do you understand how to 'balance your diet'? Have you learned new recipes, methods of cooking, or methods for storage of food that will help you plan your meals (follow by 'give examples please')? Do you understand the difference between proteins, fats and carbohydrates and foods that provide these nutrients? Health knowledge is assessed at the end of the program and one year later to determine changes to knowledge over time.
Participant Nutrition - Food Security | Food Security scores will be evaluated immediately pre-program (Week1; Time 1), after the live program (12 weeks; Time 2), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Food security will be evaluated using the 2-Item Food Security Screen. Percentage positively responding to food security questions and change over time will be completed and correlated with other outcome measures including nutritional intake, anthropometric changes, mental health and quality of life.
Awareness and access to previously unused or unknown resources | Access to resources will be evaluated immediately pre-program (Week1; Time 1), after the full program (Week 18 or 24; Time 3), and 52 weeks after the full program (Week 70 or 76; Time 4).
  Open-ended (qualitative) survey questions will assess if there are resources (ie. medical, mental health, cultural programming, recreational, food, social, etc.) that the participant faces barriers to accessing and whether their use of these resources changes with their participation in the program.
  This information will be reported in a table and will be provided to communities after the project is complete.
Attendance | Attendance is tracked throughout the program and ultimately evaluated at the end of the program (Week 18 or 24; Time 3).
  The investigators will present attendance rates as # participants/program, # attending <25%, 25- 50%, 50-75% and >75% of classes (mean attendance with range), a participant is defined as attending a program if they attended 50% or greater of the classes.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Wicklum, MD CCFP FCFP, Principal Investigator — University of Calgary; Levi Frehlich, BSc (Hons), MSc, PhD Candidate, Principal Investigator — University of Calgary
Locations (7):
- Canada (7):
  - Miskanawah, Calgary, Alberta
  - Edmonton, Edmonton, Alberta
  - Piikani First Nation, Piikani Nation, Alberta
  - Flying Dust First Nation, Flying Dust First Nation, Saskatchewan
  - Ministikwan Lake Cree Nation, Ministikwan Lake, Saskatchewan
  - Onion Lake Health Centre, Onion Lake, Saskatchewan
  - Waterhen Lake First Nation, Waterhen Lake, Saskatchewan

REFERENCES:
- [Background] Bergman RN, Stefanovski D, Buchanan TA, Sumner AE, Reynolds JC, Sebring NG, Xiang AH, Watanabe RM. A better index of body adiposity. Obesity (Silver Spring). 2011 May;19(5):1083-9. doi: 10.1038/oby.2011.38. Epub 2011 Mar 3. PMID 21372804
- [Background] Deurenberg P, Weststrate JA, Seidell JC. Body mass index as a measure of body fatness: age- and sex-specific prediction formulas. Br J Nutr. 1991 Mar;65(2):105-14. doi: 10.1079/bjn19910073. PMID 2043597
- [Background] Devlin N, Parkin D, Janssen B. Methods for Analysing and Reporting EQ-5D Data [Internet]. Cham (CH): Springer; 2020. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK565678/ PMID 33347096
- [Background] Forde C. Exercise Prescription for the Prevention and Treatment of Disease. Scoring the International Physical Activity Questionnaire (IPAQ). Trinity College Dublin, The University of Dublin. 2016. https://ugc.futurelearn.com/uploads/files/bc/c5/bcc53b14-ec1e-4d90-88e3-1568682f32ae/IPAQ_PDF.pdf
- [Background] Frehlich L, Blackstaffe A, McCormack GR. Test-Retest Reliability and Walk Score(R) Neighbourhood Walkability Comparison of an Online Perceived Neighbourhood-Specific Adaptation of the International Physical Activity Questionnaire (IPAQ). Int J Environ Res Public Health. 2019 May 30;16(11):1917. doi: 10.3390/ijerph16111917. PMID 31151210
- [Background] Halls, S.B. Body Fat Percentage: Find Out Yours. Halls.md. Body fat percentage formula from body mass index (halls.md). 2019.
- [Background] Kading ML, Hautala DS, Palombi LC, Aronson BD, Smith RC, Walls ML. Flourishing: American Indian Positive Mental Health. Soc Ment Health. 2015 Nov;5(3):203-217. doi: 10.1177/2156869315570480. Epub 2015 Feb 2. PMID 28966866
- [Background] Radandt NE, Corbridge T, Johnson DB, Kim AS, Scott JM, Coldwell SE. Validation of a Two-Item Food Security Screening Tool in a Dental Setting. J Dent Child (Chic). 2018 Sep 15;85(3):114-119. PMID 30869587
- [Background] Sallis JF, Bowles HR, Bauman A, Ainsworth BE, Bull FC, Craig CL, Sjostrom M, De Bourdeaudhuij I, Lefevre J, Matsudo V, Matsudo S, Macfarlane DJ, Gomez LF, Inoue S, Murase N, Volbekiene V, McLean G, Carr H, Heggebo LK, Tomten H, Bergman P. Neighborhood environments and physical activity among adults in 11 countries. Am J Prev Med. 2009 Jun;36(6):484-90. doi: 10.1016/j.amepre.2009.01.031. PMID 19460656
- [Background] Wicklum, S., Sampson, M., Henderson, R., Wiart, S., Perez, G., McGuire, A., Cameron, E., Willis, E., Crowshoe, L., McBrien, K. Results of a culturally relevant, physical activity-based wellness program for urban indigenous women in Alberta, Canada. International Journal of Indigenous Health. 2019; 14(2), 169-204. https://doi.org/10.32799/ijih.v14i2.31890.
- [Background] Rao DP, Dai S, Lagace C, Krewski D. Metabolic syndrome and chronic disease. Chronic Dis Inj Can. 2014 Feb;34(1):36-45. English, French. PMID 24618380
- [Background] Robinson CA, Agarwal G, Nerenberg K. Validating the CANRISK prognostic model for assessing diabetes risk in Canada's multi-ethnic population. Chronic Dis Inj Can. 2011 Dec;32(1):19-31. PMID 22153173

DOCUMENTS (1):
  • Informed Consent Form (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT05362435/ICF_000.pdf